CLINICAL TRIAL: NCT02191202
Title: Observational Study of the Impact on Quality-of-life of a Switch From a Virologically Effective Regimen to a Regimen Containing a Non-Nucleoside Reverse Transcriptase Inhibitor (QUALVI) Nevirapine (Viramune®) Clinical Phase IV
Brief Title: Impact of Switching to NNRTI-based Therapy on the Quality of Life of HIV-infected Patients With Virological Suppression
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1100.1461
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTI)
  Interventions: Drug: Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTI)

INTERVENTIONS:
Drug: Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTI)

SUMMARY:
Observational study to evaluate therapeutic switch to a NNRTI-based regimen on quality of life of HIV-positive patients

ELIGIBILITY:
Inclusion Criteria:

* NNRTI-naive patients with positive HIV serology, treated with at least triple combination therapy, with a viral load < 500 copies/ml, in whom a new treatment comprising an NNRTI is initiated for a reason other than inefficacy of treatment will be included
* Patients must read and write French

Exclusion Criteria:

* Patients in whom a new treatment is initiated because of treatment failure
* new treatment does not comprise an NNRTI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital physicians, specialized in treatment of patients infected by the HIV
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2004-06; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Changes in World Health Organization Quality of Life - HIV (WHOQOL-HIV) score | Baseline, month 1, 6 and 12

SECONDARY OUTCOMES:
Comparison of Short version of the Medical Outcomes Study Short-Form General Health Survey-36 (SF12) scores of the study population compared to the general population | Baseline, 12 months
Changes in symptom scale score | Baseline, month 1, 6 and 12
Changes in Hospital Anxiety and Depression scale (HADS) | Baseline, month 1, 6 and 12
Changes in cluster of differentiation 4 (CD4) cell count | Baseline and month 3, 6, 9, 12
Changes in viral load | Baseline and month 3, 6, 9, 12
Changes in liver function tests | Baseline and month 3, 6, 9, 12
Changes in total cholesterol | Baseline, month 6 and 12
Changes in triglycerides | Baseline, month 6 and 12
Changes in fasting blood glucose | Baseline, month 6 and 12
Changes in haemoglobin | Baseline, month 6 and 12
Changes from baseline in plasma urea | Baseline, month 12
Changes from baseline in creatinine | Baseline, month 12